CLINICAL TRIAL: NCT00438555
Title: Randomized, Controlled, Open, Comparative Intervention Study for Obesity Prevention in Children
Acronym: 4055obesityprv
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: rmc004055ctil
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2014-07

CONDITIONS: Obesity
Keywords: obesity,prevention,pediatric
MeSH Terms: conditions — Obesity

ARMS (3):
- Parent's group (Experimental): 3 months workshop of parents intervention, guided by dietician and phycologist
  Interventions: Behavioral: Parent's group
- Parents and children group (Experimental): 3 months workshops of parents and children intervention, guided by dietician and phycologist
  Interventions: Behavioral: Parents and children group
- Control group (No Intervention): control group, no intervention, medical follow up only

INTERVENTIONS:
Behavioral: Parents and children group — 3 months workshops of parents and children intervention, guided by dietician and phycologist
  Arms: Parents and children group
Behavioral: Parent's group — 3 months workshop of parents intervention, guided by dietician and phycologist
  Arms: Parent's group

SUMMARY:
Randomized, controlled, open, comparative intervention study in 270 children at risk for obesity.Patients will be randomly allocated into one of two behavior intervention groups or control group in ratio of 1:1:1.The study will consist of two main periods: an intervention period of 3 months followed by 21 months of a follow up period. During the intervention period, participants (parents or both parents and children, depending on randomization) will attend a behavior intervention program once a week, each session will last one hour and would be guided by dietician and psychologist. Follow up visits will be performed at the clinic (for participants in al 3 groups) at months 0, 3, 12 and 24.

DETAILED DESCRIPTION:
Randomized, controlled, open, comparative intervention study in 270 children at risk for obesity.

Objectives:

1. To develop an intervention program for obesity prevention in children aged 5-10 years old, who are at risk to develop obesity
2. To compare between the efficacy of two different intervention programs and a control group in preventing obesity in the short and the long term.
3. To evaluate the role and significance of including parents in an intervention program for obesity prevention.
4. To identify demographic parameters, lifestyle characteristic and biochemical markers that predict the risk of developing obesity and the response for treatment.

Randomization:

Patients will be randomly allocated into one of two intervention groups or control group in ratio of 1:1:1. Each group will contain 12-15 participants.

Intervention groups:

1. parent's group- only parents will take part at the intervention program.
2. Parents and children group- both children and parents will take part at the intervention program, in two separate sessions.

Methods:

1. The study will be consist of two main periods: an intervention period of 3 months followed by 21 months of a follow up period. During the intervention period, participants (parents or both parents and children, depending on randomization) will attend a behavior intervention program once a week, each session will last one hour and would be guided by dietician and psychologist. Follow up visits will be performed at the clinic (for participants in all 3 groups) at months 0, 3, 12 and 24.
2. Height, weight, fat mass and waist circumference will be measured at 0, 3, 12 and 24 month. Height and weight of parents will also be measured at these visits.
3. Physical examination will be performed at 0, 3, 12 and 24 month.
4. Psychological and nutritional questionnaire (depression, quality of life and self estimation) will be filled at 0, 3, 12 and 24 month.
5. Fasting blood tests for: chemistry, hematology, lipids, glucose, insulin, TSH, adiponectin, IL-6 and TNFα will be performed at 0, 3, 12 and 24 month.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-10 years old
* BMI in 85-98 percentile
* Both parents signing informed consent form

Exclusion Criteria:

* Chronic disease or chronic use of medication
* Incapability to perform all study procedure

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 248 (Actual)
Dates: Start 2006-10; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
BMI | 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, MD, Principal Investigator — Schneider Children Medical Center; Joseph Meyerovitch, Dr, MD, Principal Investigator — Schneider Children Medical Center
Locations (1):
- schneider children medical center of Israel, Petah Tikva, Israel